CLINICAL TRIAL: NCT02353923
Title: OcuStem Nutritional Supplement in Diabetic Patients With Mild to Moderate Non-proliferative Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aidan Products LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OcuStem-001
Record Dates: First submitted 2014-10-17; First posted 2015-02-03 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OcuStem Supplementation (Experimental): Twice daily supplementation with OcuStem. Subjects will take 2 capsules in the morning and 2 capsules at night for a total of 2800 mg/day of active ingredients.
  Interventions: Dietary Supplement: OcuStem Supplementation

INTERVENTIONS:
Dietary Supplement: OcuStem Supplementation — 2800 mg daily dosage of OcuStem, 2 capsules BID.

SUMMARY:
The purpose of this study is to determine whether supplementation with OcuStem, a nutritional supplement, will reduce the progression of mild to moderate diabetic retinopathy.

DETAILED DESCRIPTION:
This research study is designed to evaluate the effects of a nutritional supplement, OcuStem, on mild to moderate nonproliferative diabetic retinopathy. In this condition blood vessels in the back of the eye, an area termed the retina, are deteriorating. OcuStem contains ingredients that have previously been demonstrated in clinical trials to stimulate a type of cell, called "endothelial progenitor cells" to increase in circulation. Animal studies have shown that increasing endothelial progenitor cell numbers inhibits progression of diabetic retinopathy. The hypothesis of the study is that a 6 month course of OcuStem will reduce progression of mild to moderate diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* One or both study eyes per subject may be enrolled.
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Any one of the following will be considered to be sufficient evidence that diabetes is present:

  1. Current regular use of insulin for the treatment of diabetes
  2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
  3. Documented diabetes by ADA and/or WHO criteria.
* The study eye must meet the following:

  1. Presence of microaneurysms or at least mild non-proliferative diabetic retinopathy (level 20 or higher) on clinical exam.
  2. No presence of center-involved diabetic macular edema (DME) as evidenced by OCT central subfield thickness <250 microns(or spectral domain OCT equivalent).
  3. Visual acuity light perception or better.

Exclusion Criteria:

* A current ocular condition that, in the opinion of the investigator, visual acuity might be affected now and/or may need to be treated (e.g., DME, foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition (cataract ), epiretinal membrane or vitro-macular traction) or during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
* A history of a major ocular surgery (including vitrectomy, scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery including cataract removal anticipated within the next 4 months following enrollment.
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in Electronic-ETDRS (Early Treatment Diabetic Retinopathy Study) visual acuity testing | 0 months, 3 months, 6 months
  Electronic-ETDRS visual acuity testing at 3 meters using the Electronic Visual Acuity Tester (including protocol refraction) in each eye

SECONDARY OUTCOMES:
Change in Optical Coherence Tomography OCT (Optical Coherence Tomography) | 0 months, 3 months, 6 months
  Optical Coherence Tomography OCT on the study eye or eyes. This is to determine if there is any development of diabetic macular edema
Change in Fluorescein Angiography | 0 months, 3 months, 6 months
  Fluorescein Angiography on the study eye or eyes. This is to determine if there is any subtle evidence of diabetic changes including microaneurisms or mild macular edema.
Change in Microperimetry testing of macular function | 0 months, 3 months, 6 months
  Microperimetry testing of macular function. This non-invasive test measures retinal sensitivity to various intensities of light in a defined region of the macula
Change in Hemoglobin A1C blood levels | 0 months, 3 months, 6 months
  This is a well-established standard marker for diabetic control
Change in Blood levels of circulating endothelial progenitor cells (EPC) | 0 months, 3 months, 6 months
  Blood levels of circulating endothelial progenitor cells (EPC) as determined by CD34 levels

CONTACTS AND LOCATIONS:
Overall Officials: Shalesh Kaushal, MD, Principal Investigator — Retina Specialty Institute